CLINICAL TRIAL: NCT05067270
Title: A Study to Investigate Local Infusion Site Pain After Infusion of Excipients Across Infusion Sites and Infusion Depths
Brief Title: A Study of Infusion Site Pain After Infusion of Excipients in Participants With Type 1 Diabetes Mellitus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 18278; I8B-MC-ITTC (Other: Eli Lilly and Company); 2021-001987-18 (EudraCT Number)
Record Dates: First submitted 2021-09-28; First posted 2021-10-05 (Actual); Results first posted 2023-10-04 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2022-12

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Humalog - Insulin lispro; Citrate; Infusion Site Pain; Excipients
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Sodium Citrate; treprostinil; Magnesium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Sequence 1:Arm Region,Abdomen 6mm,Buttock,Abdomen 9mm,Thigh (Experimental): Participants had cannulas inserted into each of the designated infusion sites (6 millimeter (mm) for all the sites. Additionally for the abdominal area only, a 9 mm cannula was also inserted into the opposite side of the lower abdomen), and the first infusion site was initiated subcutaneously (SC) with 15 millimolar (mM) sodium citrate and 1 microgram per milliliter (μg/mL) treprostinil in Humalog diluent with 5 mM magnesium chloride (without insulin) solution at a basal infusion rate of 1 unit per hour (U/h). The same procedure occurred at subsequent infusion sites with an approximately 30-minute (min) interval between each initiation. Approximately 3, 6, and 9 hours after the start of the basal infusion, a bolus dose of 15 U was delivered at quick bolus speed (15 U/min) to each infusion site according to the treatment sequence with an approximately 30-minute interval between infusion sites.
  Interventions: Drug: Sodium Citrate; Drug: Treprostinil; Drug: Humalog diluent; Drug: Magnesium Chloride
- Sequence 2:Abdomen 6mm,Abdomen 9mm,Arm Region,Thigh,Buttock (Experimental): Participants had cannulas inserted into each of the designated infusion sites (6 mm for all the sites. Additionally for the abdominal area only, a 9 mm cannula was also inserted into the opposite side of the lower abdomen), and the first infusion site was initiated with 15 mM sodium citrate and 1 μg/mL treprostinil in Humalog diluent with 5 mM magnesium chloride (without insulin) solution at a basal infusion rate of 1 U/h. The same procedure occurred at subsequent infusion sites with an approximately 30-minute interval between each initiation. Approximately 3, 6, and 9 hours after the start of the basal infusion, a bolus dose of 15 U was delivered at quick bolus speed (15 U/min) to each infusion site according to the treatment sequence with an approximately 30-minute interval between infusion sites.
  Interventions: Drug: Sodium Citrate; Drug: Treprostinil; Drug: Humalog diluent; Drug: Magnesium Chloride
- Sequence 3:Abdomen 9mm,Thigh,Abdomen 6mm,Buttock,Arm Region (Experimental): Participants had cannulas inserted into each of the designated infusion sites (6 mm for all the sites. Additionally for the abdominal area only, a 9 mm cannula was also inserted into the opposite side of the lower abdomen), and the first infusion site was initiated with 15 mM sodium citrate and 1 μg/mL treprostinil in Humalog diluent with 5 mM magnesium chloride (without insulin) solution at a basal infusion rate of 1 U/h. The same procedure occurred at subsequent infusion sites with an approximately 30-minute interval between each initiation. Approximately 3, 6, and 9 hours after the start of the basal infusion, a bolus dose of 15 U was delivered at quick bolus speed (15 U/min) to each infusion site according to the treatment sequence with an approximately 30-minute interval between infusion sites.
  Interventions: Drug: Sodium Citrate; Drug: Treprostinil; Drug: Humalog diluent; Drug: Magnesium Chloride
- Sequence 4:Thigh,Buttock,Abdomen 9mm,Arm Region,Abdomen 6mm (Experimental): Participants had cannulas inserted into each of the designated infusion sites (6 mm for all the sites. Additionally for the abdominal area only, a 9 mm cannula was also inserted into the opposite side of the lower abdomen), and the first infusion site was initiated with 15 mM sodium citrate and 1 μg/mL treprostinil in Humalog diluent with 5 mM magnesium chloride (without insulin) solution at a basal infusion rate of 1 units per U/h. The same procedure occurred at subsequent infusion sites with an approximately 30-minute interval between each initiation. Approximately 3, 6, and 9 hours after the start of the basal infusion, a bolus dose of 15 U was delivered at quick bolus speed (15 U/min) to each infusion site according to the treatment sequence with an approximately 30-minute interval between infusion sites.
  Interventions: Drug: Sodium Citrate; Drug: Treprostinil; Drug: Humalog diluent; Drug: Magnesium Chloride
- Sequence 5:Buttock,Arm Region,Thigh,Abdomen 6mm,Abdomen 9mm (Experimental): Participants had cannulas inserted into each of the designated infusion sites (6 mm for all the sites. Additionally for the abdominal area only, a 9 mm cannula was also inserted into the opposite side of the lower abdomen), and the first infusion site was initiated with 15 mM sodium citrate and 1 μg/mL treprostinil in Humalog diluent with 5 mM magnesium chloride (without insulin) solution at a basal infusion rate of 1 U/h. The same procedure occurred at subsequent infusion sites with an approximately 30-minute interval between each initiation. Approximately 3, 6, and 9 hours after the start of the basal infusion, a bolus dose of 15 U was delivered at quick bolus speed (15 U/min) to each infusion site according to the treatment sequence with an approximately 30-minute interval between infusion sites.
  Interventions: Drug: Sodium Citrate; Drug: Treprostinil; Drug: Humalog diluent; Drug: Magnesium Chloride

INTERVENTIONS:
Drug: Sodium Citrate — Administered SC infusion.
Drug: Treprostinil — Administered SC infusion.
Drug: Humalog diluent — Administered SC infusion.
Drug: Magnesium Chloride — Administered SC infusion.

SUMMARY:
The main purpose of this study is to evaluate the effect of excipients sodium citrate and treprostinil without insulin on local infusion site pain in participants with type 1 diabetes mellitus (T1DM) on continuous subcutaneous insulin infusion (CSII). The study may last up to 36 days including a screening period and 3 visits.

ELIGIBILITY:
Inclusion Criteria:

* T1D for at least 1 year and continuously using insulin for at least 1 year
* Using an insulin pump for at least the last 6 months
* Have hemoglobin A1c (HbA1c) value of ≤ 9.0%
* Have a body mass index (BMI) within the range of 18.5 to 35.0 kilograms per square meter (kg/m²)
* Have medical and laboratory test results that are acceptable for the study
* Have venous access sufficient to allow for blood sampling

Exclusion Criteria:

* Hemophilia or any other bleeding disorder
* Have a pathologic tuning fork test as assessed with a Rydel-Seiffer tuning fork
* Are taking anesthetics or pain medication regularly or intermittently which could interfere with interpretation of pain scale
* Have had more than 1 episode of severe hypoglycemia (defined as requiring assistance due to neurologically disabling hypoglycemia) within the last 90 days prior to screening
* Have had more than 1 emergency room visit or hospitalization due to poor glucose control (hyperglycemia or diabetic ketoacidosis) within the last 6 months prior to screening
* Have any hypersensitivity or allergy to any of the diluents or excipients used in this trial
* Have or used to have health problems or medical test results that, in the opinion of the doctor, could make it unsafe to participate, or could interfere with understanding the results of the study
* Have participated, within the last 30 days, in a clinical trial involving an investigational product
* Have used or are currently using Lyumjev® as part of their standard insulin therapy

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-10-22 (Actual); Primary Completion 2021-12-06 (Actual); Study Completion 2021-12-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (2):
- Germany (2):
  - Profil Institut für Stoffwechselforschung, Neuss, North Rhine-Westphalia
  - Profil Mainz, Mainz

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ignaut D, Fukuda T, Bandi R, Ermer M, Stoffel MS, Zijlstra E, Paavola C. An Investigation Into Local Infusion Site Pain After Infusion of Ultra Rapid Lispro Excipients Across Sites and Depths. J Diabetes Sci Technol. 2024 Jul;18(4):920-929. doi: 10.1177/19322968221135217. Epub 2022 Nov 3. PMID 36326260

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were randomly assigned to 1 of 5 infusion site sequence below and received the study treatment in each period. Cannulas were inserted into each of the designated infusion sites (6 millimeter (mm) for all the sites. Additionally for the abdominal area only, a 9 mm cannula was also inserted into the opposite side of the lower abdomen).
Groups:
- Sequence 1:Arm Region,Abdomen 6mm,Buttock,Abdomen 9mm,Thigh: Participants received 15 millimolar (mM) sodium citrate and 1 microgram per milliliter (μg/mL) treprostinil in Humalog diluent with 5 mM magnesium chloride (without insulin) solution as subcutaneous (SC) infusion at the first infusion site at a basal infusion rate of 1 unit per hour (U/h). The same procedure occurred at subsequent infusion sites with an approximately 30-minute (min) interval between each initiation. Approximately 3, 6, and 9 hours after the start of the basal infusion, a bolus dose of 15 U was delivered at quick bolus speed (15 U/min) to each infusion site according to the treatment sequence with an approximately 30-minute interval between infusion sites.
  Period 1: Arm region; Period 2: Abdomen 6mm; Period 3: Buttock; Period 4: Abdomen 9mm; Period 5: Thigh.
- Sequence 2:Abdomen 6mm,Abdomen 9mm,Arm Region,Thigh,Buttock: Participants received 15 mM sodium citrate and 1 μg/mL treprostinil in Humalog diluent with 5 mM magnesium chloride (without insulin) solution as SC infusion at the first infusion site at a basal infusion rate of 1 U/h. The same procedure occurred at subsequent infusion sites with an approximately 30-minute interval between each initiation. Approximately 3, 6, and 9 hours after the start of the basal infusion, a bolus dose of 15 U was delivered at quick bolus speed (15 U/min) to each infusion site according to the treatment sequence with an approximately 30-minute interval between infusion sites.
  Period 1: Abdomen 6mm; Period 2: Abdomen 9mm; Period 3: Arm region; Period 4: Thigh; Period 5: Buttock.
- Sequence 3:Abdomen 9mm,Thigh,Abdomen 6mm,Buttock,Arm Region: Participants received 15 mM sodium citrate and 1 μg/mL treprostinil in Humalog diluent with 5 mM magnesium chloride (without insulin) solution as SC infusion at the first infusion site at a basal infusion rate of 1 U/h. The same procedure occurred at subsequent infusion sites with an approximately 30-minute interval between each initiation. Approximately 3, 6, and 9 hours after the start of the basal infusion, a bolus dose of 15 U was delivered at quick bolus speed (15 U/min) to each infusion site according to the treatment sequence with an approximately 30-minute interval between infusion sites.
  Period 1: Abdomen 9mm; Period 2: Thigh; Period 3: Abdomen 6mm; Period 4: Buttock; Period 5: Arm region.
- Sequence 4:Thigh,Buttock,Abdomen 9mm,Arm Region,Abdomen 6mm: Participants received 15 mM sodium citrate and 1 μg/mL treprostinil in Humalog diluent with 5 mM magnesium chloride (without insulin) solution as SC infusion at the first infusion site at a basal infusion rate of 1 U/h. The same procedure occurred at subsequent infusion sites with an approximately 30-minute interval between each initiation. Approximately 3, 6, and 9 hours after the start of the basal infusion, a bolus dose of 15 U was delivered at quick bolus speed (15 U/min) to each infusion site according to the treatment sequence with an approximately 30-minute interval between infusion sites.
  Period 1: Thigh; Period 2: Buttock; Period 3: Abdomen 9mm; Period 4: Arm Region; Period 5: Abdomen 6mm.
- Sequence 5:Buttock,Arm Region,Thigh,Abdomen 6mm,Abdomen 9mm: Participants received 15 mM sodium citrate and 1 μg/mL treprostinil in Humalog diluent with 5 mM magnesium chloride (without insulin) solution as SC infusion at the first infusion site at a basal infusion rate of 1 U/h. The same procedure occurred at subsequent infusion sites with an approximately 30-minute interval between each initiation. Approximately 3, 6, and 9 hours after the start of the basal infusion, a bolus dose of 15 U was delivered at quick bolus speed (15 U/min) to each infusion site according to the treatment sequence with an approximately 30-minute interval between infusion sites.
  Period 1: Buttock; Period 2: Arm region; Period 3: Thigh; Period 4: Abdomen 6mm; Period 5: Abdomen 9mm.
Period: Period 1
Arm/Group | Sequence 1:Arm Region,Abdomen 6mm,Buttock,Abdomen 9mm,Thigh | Sequence 2:Abdomen 6mm,Abdomen 9mm,Arm Region,Thigh,Buttock | Sequence 3:Abdomen 9mm,Thigh,Abdomen 6mm,Buttock,Arm Region | Sequence 4:Thigh,Buttock,Abdomen 9mm,Arm Region,Abdomen 6mm | Sequence 5:Buttock,Arm Region,Thigh,Abdomen 6mm,Abdomen 9mm
Started | 8 | 8 | 8 | 8 | 8
Received At Least One Infusion | 8 | 8 | 8 | 8 | 8
Completed | 8 | 8 | 8 | 8 | 8
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Period 2
Arm/Group | Sequence 1:Arm Region,Abdomen 6mm,Buttock,Abdomen 9mm,Thigh | Sequence 2:Abdomen 6mm,Abdomen 9mm,Arm Region,Thigh,Buttock | Sequence 3:Abdomen 9mm,Thigh,Abdomen 6mm,Buttock,Arm Region | Sequence 4:Thigh,Buttock,Abdomen 9mm,Arm Region,Abdomen 6mm | Sequence 5:Buttock,Arm Region,Thigh,Abdomen 6mm,Abdomen 9mm
Started | 8 | 8 | 8 | 8 | 8
Received At Least One Infusion | 8 | 8 | 8 | 8 | 8
Completed | 8 | 8 | 8 | 8 | 8
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Period 3
Arm/Group | Sequence 1:Arm Region,Abdomen 6mm,Buttock,Abdomen 9mm,Thigh | Sequence 2:Abdomen 6mm,Abdomen 9mm,Arm Region,Thigh,Buttock | Sequence 3:Abdomen 9mm,Thigh,Abdomen 6mm,Buttock,Arm Region | Sequence 4:Thigh,Buttock,Abdomen 9mm,Arm Region,Abdomen 6mm | Sequence 5:Buttock,Arm Region,Thigh,Abdomen 6mm,Abdomen 9mm
Started | 8 | 8 | 8 | 8 | 8
Received At Least One Infusion | 8 | 8 | 8 | 8 | 8
Completed | 8 | 8 | 8 | 8 | 8
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Period 4
Arm/Group | Sequence 1:Arm Region,Abdomen 6mm,Buttock,Abdomen 9mm,Thigh | Sequence 2:Abdomen 6mm,Abdomen 9mm,Arm Region,Thigh,Buttock | Sequence 3:Abdomen 9mm,Thigh,Abdomen 6mm,Buttock,Arm Region | Sequence 4:Thigh,Buttock,Abdomen 9mm,Arm Region,Abdomen 6mm | Sequence 5:Buttock,Arm Region,Thigh,Abdomen 6mm,Abdomen 9mm
Started | 8 | 8 | 8 | 8 | 8
Received At Least One Infusion | 8 | 8 | 8 | 8 | 8
Completed | 8 | 8 | 8 | 8 | 8
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Period 5
Arm/Group | Sequence 1:Arm Region,Abdomen 6mm,Buttock,Abdomen 9mm,Thigh | Sequence 2:Abdomen 6mm,Abdomen 9mm,Arm Region,Thigh,Buttock | Sequence 3:Abdomen 9mm,Thigh,Abdomen 6mm,Buttock,Arm Region | Sequence 4:Thigh,Buttock,Abdomen 9mm,Arm Region,Abdomen 6mm | Sequence 5:Buttock,Arm Region,Thigh,Abdomen 6mm,Abdomen 9mm
Started | 8 | 8 | 8 | 8 | 8
Received At Least One Infusion | 8 | 8 | 8 | 8 | 8
Completed | 8 | 8 | 8 | 8 | 8
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received at least one Infusion.
Groups:
- Overall: Participants received 15 mM sodium citrate and 1 μg/mL treprostinil in humalog diluent with 5 mM magnesium chloride (without insulin) as SC infusion.
  Six mm cannula was inserted into each of the designated areas (arm, abdomen, thigh, and buttock). At the abdominal area only, a 9 mm cannula was also inserted into the opposite side of the lower abdomen.
Arm/Group | Overall
Number analyzed (Participants) | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.5 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 30
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 40
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Germany | 40

OUTCOME MEASURES:

1. Primary Outcome: Visual Analog Scale (VAS) Pain Score in the Abdominal, Arm, Thigh, and Buttock Areas
Description: The Infusion site pain VAS score is a participant administered single item scale designed to measure pain using a 0-100 millimeter (mm) horizontal VAS. Overall severity of participant's pain is indicated by placing a single mark on the horizontal 100 mm scale from 0 mm (no pain) to 100 mm (worst imaginable pain).
Time Frame: Day 1: 1 min post bolus.
Population: All participants who received at least one infusion and had VAS pain scores.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: millimeter
Groups:
- Treatment Given to Arm Region: Participants received 15 mM sodium citrate and 1 μg/mL treprostinil in humalog diluent with 5 mM magnesium chloride (without insulin) as SC infusion to the arm.
- Treatment Given to Thigh: Participants received 15 mM sodium citrate and 1 μg/mL treprostinil in humalog diluent with 5 mM magnesium chloride (without insulin) as SC infusion to thigh.
- Treatment Given to Abdomen (6 mm): Participants received 15 mM sodium citrate and 1 μg/mL treprostinil in humalog diluent with 5 mM magnesium chloride (without insulin) as SC infusion through a 6mm cannula to the abdomen.
- Treatment Given to Abdomen (9 mm): Participants received 15 mM sodium citrate and 1 μg/mL treprostinil in humalog diluent with 5 mM magnesium chloride (without insulin) as SC infusion through a 9 mm cannula to the abdomen.
- Treatment Given to Buttock: Participants received 15 mM sodium citrate and 1 μg/mL treprostinil in humalog diluent with 5 mM magnesium chloride (without insulin) as SC infusion to the buttock.
Arm/Group | Treatment Given to Arm Region | Treatment Given to Thigh | Treatment Given to Abdomen (6 mm) | Treatment Given to Abdomen (9 mm) | Treatment Given to Buttock
Number analyzed (Participants) | 38 | 37 | 39 | 40 | 39
millimeter
  1 min post bolus (Bolus time: 3 hours) | 3.4 (182) | 2.0 (119) | 1.8 (112) | 1.9 (119) | 2.4 (167)
  1 min post bolus (Bolus time: 6 hours): number analyzed (Participants) | 38 | 36 | 39 | 40 | 39
  1 min post bolus (Bolus time: 6 hours) | 3.7 (164) | 2.6 (137) | 2.3 (151) | 2.0 (113) | 3.3 (161)
  1 min post bolus (Bolus time: 9 hours): number analyzed (Participants) | 38 | 36 | 39 | 40 | 39
  1 min post bolus (Bolus time: 9 hours) | 4.8 (211) | 3.4 (155) | 2.5 (141) | 2.4 (141) | 3.8 (196)
Statistical Analysis 1: Comparison: Treatment Given to Arm Region vs Treatment Given to Thigh; 1 min post bolus (Bolus time: 3 hours); Test type: Other; Geometric Least Squares Mean Ratio = 1.77, 95% CI 2-sided [1.30 to 2.40]
Statistical Analysis 2: Comparison: Treatment Given to Arm Region vs Treatment Given to Abdomen (6 mm); 1 min post bolus (Bolus time: 3 hours); Test type: Other; Geometric Least Squares Mean Ratio = 1.91, 95% CI 2-sided [1.42 to 2.59]
Statistical Analysis 3: Comparison: Treatment Given to Arm Region vs Treatment Given to Abdomen (9 mm); 1 min post bolus (Bolus time: 3 hours); Test type: Other; Geometric Least Squares Mean Ratio = 1.84, 95% CI 2-sided [1.37 to 2.49]
Statistical Analysis 4: Comparison: Treatment Given to Arm Region vs Treatment Given to Buttock; 1 min post bolus (Bolus time: 3 hours); Test type: Other; Geometric Least Squares Mean Ratio = 1.42, 95% CI 2-sided [1.05 to 1.92]
Statistical Analysis 5: Comparison: Treatment Given to Thigh vs Treatment Given to Abdomen (6 mm); 1 min post bolus (Bolus time: 3 hours); Test type: Other; Geometric Least Squares Mean Ratio = 1.08, 95% CI 2-sided [0.80 to 1.46]
Statistical Analysis 6: Comparison: Treatment Given to Thigh vs Treatment Given to Abdomen (9 mm); 1 min post bolus (Bolus time: 3 hours); Test type: Other; Geometric Least Squares Mean Ratio = 1.04, 95% CI 2-sided [0.77 to 1.41]
Statistical Analysis 7: Comparison: Treatment Given to Thigh vs Treatment Given to Buttock; 1 min post bolus (Bolus time: 3 hours); Test type: Other; Geometric Least Squares Mean Ratio = 0.80, 95% CI 2-sided [0.59 to 1.08]
Statistical Analysis 8: Comparison: Treatment Given to Abdomen (6 mm) vs Treatment Given to Abdomen (9 mm); 1 min post bolus (Bolus time: 3 hours); Test type: Other; Geometric Least Squares Mean Ratio = 0.96, 95% CI 2-sided [0.72 to 1.30]
Statistical Analysis 9: Comparison: Treatment Given to Abdomen (6 mm) vs Treatment Given to Buttock; 1 min post bolus (Bolus time: 3 hours); Test type: Other; Geometric Least Squares Mean Ratio = 0.74, 95% CI 2-sided [0.55 to 1.00]
Statistical Analysis 10: Comparison: Treatment Given to Abdomen (9 mm) vs Treatment Given to Buttock; 1 min post bolus (Bolus time: 3 hours); Test type: Other; Geometric Least Squares Mean Ratio = 0.77, 95% CI 2-sided [0.57 to 1.04]
Statistical Analysis 11: Comparison: Treatment Given to Arm Region vs Treatment Given to Thigh; 1 min post bolus (Bolus time: 6 hours); Test type: Other; Geometric Least Squares Mean Ratio = 1.49, 95% CI 2-sided [1.09 to 2.02]
Statistical Analysis 12: Comparison: Treatment Given to Arm Region vs Treatment Given to Abdomen (6 mm); 1 min post bolus (Bolus time: 6 hours); Test type: Other; Geometric Least Squares Mean Ratio = 1.68, 95% CI 2-sided [1.25 to 2.28]
Statistical Analysis 13: Comparison: Treatment Given to Arm Region vs Treatment Given to Abdomen (9 mm); 1 min post bolus (Bolus time: 6 hours); Test type: Other; Geometric Least Squares Mean Ratio = 1.84, 95% CI 2-sided [1.36 to 2.48]
Statistical Analysis 14: Comparison: Treatment Given to Arm Region vs Treatment Given to Buttock; 1 min post bolus (Bolus time: 6 hours); Test type: Other; Geometric Least Squares Mean Ratio = 1.16, 95% CI 2-sided [0.85 to 1.56]
Statistical Analysis 15: Comparison: Treatment Given to Thigh vs Treatment Given to Abdomen (6 mm); 1 min post bolus (Bolus time: 6 hours); Test type: Other; Geometric Least Squares Mean Ratio = 1.13, 95% CI 2-sided [0.83 to 1.54]
Statistical Analysis 16: Comparison: Treatment Given to Thigh vs Treatment Given to Abdomen (9 mm); 1 min post bolus (Bolus time: 6 hours); Test type: Other; Geometric Least Squares Mean Ratio = 1.24, 95% CI 2-sided [0.91 to 1.68]
Statistical Analysis 17: Comparison: Treatment Given to Thigh vs Treatment Given to Buttock; 1 min post bolus (Bolus time: 6 hours); Test type: Other; Geometric Least Squares Mean Ratio = 0.78, 95% CI 2-sided [0.57 to 1.05]
Statistical Analysis 18: Comparison: Treatment Given to Abdomen (6 mm) vs Treatment Given to Abdomen (9 mm); 1 min post bolus (Bolus time: 6 hours); Test type: Other; Geometric Least Squares Mean Ratio = 1.09, 95% CI 2-sided [0.81 to 1.47]
Statistical Analysis 19: Comparison: Treatment Given to Abdomen (6 mm) vs Treatment Given to Buttock; 1 min post bolus (Bolus time: 6 hours); Test type: Other; Geometric Least Squares Mean Ratio = 0.69, 95% CI 2-sided [0.51 to 0.93]
Statistical Analysis 20: Comparison: Treatment Given to Abdomen (9 mm) vs Treatment Given to Buttock; 1 min post bolus (Bolus time: 6 hours); Test type: Other; Geometric Least Squares Mean Ratio = 0.63, 95% CI 2-sided [0.47 to 0.85]
Statistical Analysis 21: Comparison: Treatment Given to Arm Region vs Treatment Given to Thigh; 1 min post bolus (Bolus time: 9 hours); Test type: Other; Geometric Least Squares Mean Ratio = 1.49, 95% CI 2-sided [1.10 to 2.03]
Statistical Analysis 22: Comparison: Treatment Given to Arm Region vs Treatment Given to Abdomen (6 mm); 1 min post bolus (Bolus time: 9 hours); Test type: Other; Geometric Least Squares Mean Ratio = 1.96, 95% CI 2-sided [1.45 to 2.65]
Statistical Analysis 23: Comparison: Treatment Given to Arm Region vs Treatment Given to Abdomen (9 mm); 1 min post bolus (Bolus time: 9 hours); Test type: Other; Geometric Least Squares Mean Ratio = 2.03, 95% CI 2-sided [1.50 to 2.74]
Statistical Analysis 24: Comparison: Treatment Given to Arm Region vs Treatment Given to Buttock; 1 min post bolus (Bolus time: 9 hours); Test type: Other; Geometric Least Squares Mean Ratio = 1.25, 95% CI 2-sided [0.93 to 1.69]
Statistical Analysis 25: Comparison: Treatment Given to Thigh vs Treatment Given to Abdomen (6 mm); 1 min post bolus (Bolus time: 9 hours); Test type: Other; Geometric Least Squares Mean Ratio = 1.31, 95% CI 2-sided [0.97 to 1.78]
Statistical Analysis 26: Comparison: Treatment Given to Thigh vs Treatment Given to Abdomen (9 mm); 1 min post bolus (Bolus time: 9 hours); Test type: Other; Geometric Least Squares Mean Ratio = 1.36, 95% CI 2-sided [1.01 to 1.84]
Statistical Analysis 27: Comparison: Treatment Given to Thigh vs Treatment Given to Buttock; 1 min post bolus (Bolus time: 9 hours); Test type: Other; Geometric Least Squares Mean Ratio = 0.84, 95% CI 2-sided [0.62 to 1.14]
Statistical Analysis 28: Comparison: Treatment Given to Abdomen (6 mm) vs Treatment Given to Abdomen (9 mm); 1 min post bolus (Bolus time: 9 hours); Test type: Other; Geometric Least Squares Mean Ratio = 1.04, 95% CI 2-sided [0.77 to 1.40]
Statistical Analysis 29: Comparison: Treatment Given to Abdomen (6 mm) vs Treatment Given to Buttock; 1 min post bolus (Bolus time: 9 hours); Test type: Other; Geometric Least Squares Mean Ratio = 0.64, 95% CI 2-sided [0.47 to 0.86]
Statistical Analysis 30: Comparison: Treatment Given to Abdomen (9 mm) vs Treatment Given to Buttock; 1 min post bolus (Bolus time: 9 hours); Test type: Other; Geometric Least Squares Mean Ratio = 0.62, 95% CI 2-sided [0.46 to 0.83]

ADVERSE EVENTS:
Time Frame: Up to 9 days
Description: All participants who received at least one infusion. As per the Protocol, adverse events were analyzed by infusion site locations.
Groups:
- Treatment Given to Arm Region: Participants who received 15 mM sodium citrate and 1 μg/mL treprostinil in humalog diluent with 5 mM magnesium chloride (without insulin) as SC infusion to the arm region.
Arm/Group | Treatment Given to Arm Region | Treatment Given to Thigh | Treatment Given to Abdomen (6 mm) | Treatment Given to Abdomen (9 mm) | Treatment Given to Buttock
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/40 | 0/40 | 0/40 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40 | 0/40 | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 5/40 | 9/40 | 4/40 | 4/40 | 3/40
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Given to Arm Region (N=40) | Treatment Given to Thigh (N=40) | Treatment Given to Abdomen (6 mm) (N=40) | Treatment Given to Abdomen (9 mm) (N=40) | Treatment Given to Buttock (N=40)
Infusion site reaction (General disorders) | 5 (5) | 9 (9) | 4 (4) | 4 (4) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2021-10-14): https://cdn.clinicaltrials.gov/large-docs/70/NCT05067270/Prot_000.pdf
  • Statistical Analysis Plan (2022-02-02): https://cdn.clinicaltrials.gov/large-docs/70/NCT05067270/SAP_001.pdf